CLINICAL TRIAL: NCT02781701
Title: Tongue Protrusion Force: A Pilot Study
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Sponsor: Weill Medical College of Cornell University (Other)
Collaborators: Cornell University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1602017027
Record Dates: First submitted 2016-05-19; First posted 2016-05-24 (Estimated); Last update posted 2022-02-08 (Actual); Status verified 2022-01

CONDITIONS: Obstructive Sleep Apnea (OSA)
MeSH Terms: conditions — Sleep Apnea, Obstructive

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (1):
- Tongue Trainer (Experimental): The strength of participants tongue will be measured and participants will be shown how to perform tongue training exercises using a special device. Participants will be given instructions on how to perform a workout for the tongue. Each day once in the morning (am) and once in the afternoon/evening (pm), participants will train with the device and have a "tongue workout" that lasts about 10 minutes.
  Therefore, participants will work out about 20 minutes a day for 6 weeks.
  Interventions: Device: Tongue Trainer

INTERVENTIONS:
Device: Tongue Trainer — The strength of participants tongue will be measured and participants will be shown how to perform tongue training exercises using a special device. Participants will be given instructions on how to perform a workout for the tongue. Each day once in the morning (am) and once in the afternoon/evening (pm), participants will train with the device and have a "tongue workout" that lasts about 10 minutes.
  Therefore, participants will work out about 20 minutes a day for 6 weeks.

SUMMARY:
From Weill Cornell Medical College Center for Sleep Medicine, the investigators will recruit patients (N = 25) with previously documented moderate to severe OSA. They will receive an all-night in-home sleep study to document the severity of their OSA immediately before starting the training regimen. Scales and questionnaires measuring sleepiness, snoring, fatigue, and insomnia will be administered prior to starting the training and repeated after six weeks of training. Subjects may be removed from the study due to failing to adhere to the training regimen at anytime via remote data monitoring. The principal measure of the efficacy of the treatment will be the change in RDI, the number of abnormal breathing events per hour of sleep.

DETAILED DESCRIPTION:
Obstructive sleep apnea (OSA) is a condition characterized by temporary diminutions or cessations of breathing caused by repetitive collapse of the upper airway (UA) during sleep (1). OSA is a common disorder associated with abnormalities in pharyngeal anatomy and physiology in which the muscles of the airway, which normally relax during sleep, fail to provide sufficient dilatory force to balance the contractive force from inspiratory activity (2). This force imbalance serves to either partially or completely collapse the UA, thereby preventing sufficient air from reaching the lungs. These pauses in breathing lead to blood oxygen desaturation and induce neurological arousal resulting in sleep disruption and fragmentation. The cycle of airway collapse and arousal can repeat hundreds of times per night (1). According to the National Sleep Foundation, OSA affects 18-22 million Americans, 80% of whom are undiagnosed. OSA is more prevalent among overweight and older individuals and those with reduced muscle tone, skeletal anomalies such as micrognathia or retrognathia, and airways crowded by redundant or enlarged soft tissue structures.

OSA is associated with significant physiological and psychological problems. OSA results in excessive daytime sleepiness, fatigue, memory impairment, and reduced reaction time, increasing the risk for motor vehicle (3) and workplace (4) accidents. In addition, OSA sufferers face increased cardiovascular risk including hypertension, heart disease, and stroke (5). OSA has even recently been linked to increased cancer incidence (6) and mortality (7), presumably through hypoxia-induced angiogenesis.

On the morning of December 1, 2013, a Metro-North passenger train derailed in the Bronx. The accident killed 4 passengers, injured 61, and caused $9 million worth of damage. Investigators determined human error was to blame: the train engineer admitted that before reaching the curve he had "gone into a daze," allowing the train to travel at three times the posted speed limit (8). A medical examination conducted after the accident diagnosed the train engineer with OSA, which hampered his ability to fully adjust his sleep patterns to the morning shift he had begun working just two weeks prior to the accident (9).

The Harvard Medical School released a report in 2010 entitled, "The Price of Fatigue: The Surprising Economic Costs of Unmanaged Sleep Apnea," in which it estimated the annual economic cost of moderate to severe OSA in the United States to be $65-165B (compared to $60B for drunk driving and $150B for not wearing seatbelts), including $10-40B in OSA-related traffic accidents and $5-20B in OSA-related workplace accidents (10).

Existing treatments for OSA include lifestyle modifications (11) such as weight loss, position restriction, and avoidance of muscle relaxants such as alcohol and benzodiazepine drugs. Oral appliances including mandibular advancement devices and tongue retaining devices have been increasingly employed. OSA is also treated through surgery, including tonsillectomy and uvulopalatopharyngeoplasty (UPPP) to reduce tissue crowding of the UA lumen, genioglossal advancement, and maxillomandibular advancement. The most widespread and generally effective treatment for OSA, however, remains the use of various devices for maintaining positive airway pressure (PAP) such as Continuous Positive Airway Pressure (CPAP), BiLevel Positive Airway Pressure (BiPAP), and Autotitrating (AutoPAP) devices.

CPAP and related treatments are both costly and cumbersome. 40-60% of patients prescribed CPAP fail to adhere to the treatment (12; 13; 14). Patients cite comfort and lifestyle factors (sensation of claustrophobia, dry mouth, ill-fitting mask, and lack of portability of the system precluding use during travel) as reasons for abandoning treatment (15; 16). Benign Prostatic Hypertrophy (BPH), with accompanying nocturia, has also been associated with noncompliance with CPAP among older men (17). Poor compliance with CPAP is prompting the search for alternative forms of treatment for OSA.

The Genioglossus (GG), which makes up most of the body of the tongue, is the major muscle responsible for protruding the tongue and is the major UA dilator that opposes collapsing force in the pharynx upon inspiration. Reduced UA dilator force in sleep is posited to contribute to the collapse of the pharynx in OSA (Schwartz 2001). A number of controlled studies have demonstrated that strengthening the GG can result in clinically significant reductions of OSA severity.

In a randomized controlled trial (RCT) of OSA patients (18), a group that performed oropharyngeal exercises for 30 minutes a day for three months reduced the average apnea hypopnea index (AHI, the number of apnea and hypopnea events per hour of sleep) by almost 35% (22.4 to 14.7, P < 0.05). The exercises consisted of isometric and isotonic exercises involving the tongue. Another RCT (19) designed to increase UA dilator muscle strength demonstrated that playing the didgeridoo (an aboriginal wind instrument) six times per week for an average of 25 minutes per day over four months decreased average AHI by almost 50% (22.3 to 11.6, P < 0.01). Electrical stimulation of the hypoglossal nerve (which innervates the GG) also promotes UA patency during sleep. Hypoglossal stimulation reduced UA resistance in both healthy persons and subjects with OSA and reduced AHI in OSA subjects by over 50% (20).

II. Aims

The investigators assert that training the GG muscle while awake will serve to dilate the pharyngeal pathway - restriction of which results in obstructive apnea - during sleep. If confirmed, the investigators will have developed an effective behavioral treatment for OSA. The investigators anticipate it being an attractive alternative for OSA patients who are unable to acclimate to CPAP or adhere to its use for comfort or lifestyle reasons.

This IRB approved clinical study is designed to determine both an effective training regimen to increase GG muscle strength as well as obtain preliminary data on the effect of tongue protrusive force training (TPFT) on OSA. In this study, the investigators will use subjects with moderate to severe OSA. OSA severity will be assessed with a sleep study conducted prior to beginning the training regimen. After six weeks of daily training, OSA severity will be measured again with a follow-up sleep study.

ELIGIBILITY:
Inclusion Criteria:

1. Age: 21 to 70
2. At home confirmation of moderate to severe OSA (AHI 15-60)
3. BMI less than or equal to 35
4. Not currently on a weight loss plan and no intention of beginning a weight loss regimen during the duration of the study
5. If not currently treated for OSA (AHI 15-20), not planning on starting treatment for OSA during the duration of the study
6. Willing to have a diagnostic sleep study before the training
7. Willing to have a diagnostic sleep study after the training
8. Willing to perform tongue training exercises twice daily for 6 weeks
9. Willing to keep a sleep diary

Exclusion Criteria:

1. Dental problems, e.g., less than a full complement of front teeth, loose front teeth, brittle teeth, by history
2. Temporomandibular joint (TMJ) disorder by history
3. Jaw, neck, or facial muscle pain or discomfort by history
4. Consumes more than one alcoholic beverage per day and unwilling to reduce alcohol consumption to no more than one alcoholic beverage per day (muscle relaxant)
5. On benzodiazepine medication (or specific muscle relaxant)
6. Sleeps less than 5 hours per night on average (sleep deprivation can weaken UA)
7. Pregnant
8. Has had an upper airway surgical procedure for sleep apnea below the level of the nasopharynx
9. Non-English speaker or illiterate

Ages: 21 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2017-01 (Actual); Primary Completion 2021-12 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
RDI | Six weeks
  RDI (the sum of apneas, hypopneas, and milder, more subtle sleep disruptions known as respiratory effort related arousals, or RERAs, that can still lead to sleep fragmentation).

SECONDARY OUTCOMES:
TPFmax | Six Weeks
  The investigators will be monitoring the tongue protrusion force max each day for six weeks to see what changes, if any occur.
AHI | Six Weeks
  The investigators will measure AHI during the pre-screen and post screen to see what changes, if any, occur due to the six weeks of tongue training.
dur50% | Six weeks
  To determine if regular exercise of the GG muscle increases the maximum tongue protrusive force (TPFmax) and increases the duration over which the tongue is capable of exerting sub-maximal (threshold of 50% of baseline TPFmax) protrusive force (dur50%).

CONTACTS AND LOCATIONS:
Overall Officials: Matthew Ebben, Ph. D., Principal Investigator — Weill Medical College of Cornell University
Locations (1):
- Weill Cornell Medical College Center for Sleep, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No
There is no plan to make IPD available.

REFERENCES:
- [Background] Shepherd KL, Jensen CM, Maddison KJ, Hillman DR, Eastwood PR. Relationship between upper airway and inspiratory pump muscle force in obstructive sleep apnea. Chest. 2006 Dec;130(6):1757-64. doi: 10.1378/chest.130.6.1757. PMID 17166993
- [Background] Malhotra A, Huang Y, Fogel RB, Pillar G, Edwards JK, Kikinis R, Loring SH, White DP. The male predisposition to pharyngeal collapse: importance of airway length. Am J Respir Crit Care Med. 2002 Nov 15;166(10):1388-95. doi: 10.1164/rccm.2112072. PMID 12421747
- [Background] Eastwood PR, Barnes M, Walsh JH, Maddison KJ, Hee G, Schwartz AR, Smith PL, Malhotra A, McEvoy RD, Wheatley JR, O'Donoghue FJ, Rochford PD, Churchward T, Campbell MC, Palme CE, Robinson S, Goding GS, Eckert DJ, Jordan AS, Catcheside PG, Tyler L, Antic NA, Worsnop CJ, Kezirian EJ, Hillman DR. Treating obstructive sleep apnea with hypoglossal nerve stimulation. Sleep. 2011 Nov 1;34(11):1479-86. doi: 10.5665/sleep.1380. PMID 22043118
- [Background] Peppard PE, Young T, Palta M, Skatrud J. Prospective study of the association between sleep-disordered breathing and hypertension. N Engl J Med. 2000 May 11;342(19):1378-84. doi: 10.1056/NEJM200005113421901. PMID 10805822
- [Background] Yaggi HK, Concato J, Kernan WN, Lichtman JH, Brass LM, Mohsenin V. Obstructive sleep apnea as a risk factor for stroke and death. N Engl J Med. 2005 Nov 10;353(19):2034-41. doi: 10.1056/NEJMoa043104. PMID 16282178
- [Background] Eikermann M, Jordan AS, Chamberlin NL, Gautam S, Wellman A, Lo YL, White DP, Malhotra A. The influence of aging on pharyngeal collapsibility during sleep. Chest. 2007 Jun;131(6):1702-9. doi: 10.1378/chest.06-2653. Epub 2007 Apr 5. PMID 17413053
- [Background] Campos-Rodriguez F, Martinez-Garcia MA, Martinez M, Duran-Cantolla J, Pena Mde L, Masdeu MJ, Gonzalez M, Campo Fd, Gallego I, Marin JM, Barbe F, Montserrat JM, Farre R; Spanish Sleep Network. Association between obstructive sleep apnea and cancer incidence in a large multicenter Spanish cohort. Am J Respir Crit Care Med. 2013 Jan 1;187(1):99-105. doi: 10.1164/rccm.201209-1671OC. Epub 2012 Nov 15. PMID 23155146
- [Background] Martinez-Garcia MA, Campos-Rodriguez F, Duran-Cantolla J, de la Pena M, Masdeu MJ, Gonzalez M, Del Campo F, Serra PC, Valero-Sanchez I, Ferrer MJ, Marin JM, Barbe F, Martinez M, Farre R, Montserrat JM; Spanish Sleep Network. Obstructive sleep apnea is associated with cancer mortality in younger patients. Sleep Med. 2014 Jul;15(7):742-8. doi: 10.1016/j.sleep.2014.01.020. Epub 2014 May 15. PMID 24907033
- [Background] Busetto L, Enzi G, Inelmen EM, Costa G, Negrin V, Sergi G, Vianello A. Obstructive sleep apnea syndrome in morbid obesity: effects of intragastric balloon. Chest. 2005 Aug;128(2):618-23. doi: 10.1378/chest.128.2.618. PMID 16100146
- [Background] Wolkove N, Baltzan M, Kamel H, Dabrusin R, Palayew M. Long-term compliance with continuous positive airway pressure in patients with obstructive sleep apnea. Can Respir J. 2008 Oct;15(7):365-9. doi: 10.1155/2008/534372. PMID 18949106
- [Background] Wang Y, Gao W, Sun M, Chen B. Adherence to CPAP in patients with obstructive sleep apnea in a Chinese population. Respir Care. 2012 Feb;57(2):238-43. doi: 10.4187/respcare.01136. Epub 2011 Jul 12. PMID 21762553
- [Background] Weaver TE, Kribbs NB, Pack AI, Kline LR, Chugh DK, Maislin G, Smith PL, Schwartz AR, Schubert NM, Gillen KA, Dinges DF. Night-to-night variability in CPAP use over the first three months of treatment. Sleep. 1997 Apr;20(4):278-83. doi: 10.1093/sleep/20.4.278. PMID 9231953
- [Background] Weaver TE, Sawyer AM. Adherence to continuous positive airway pressure treatment for obstructive sleep apnoea: implications for future interventions. Indian J Med Res. 2010 Feb;131:245-58. PMID 20308750
- [Background] Russo-Magno P, O'Brien A, Panciera T, Rounds S. Compliance with CPAP therapy in older men with obstructive sleep apnea. J Am Geriatr Soc. 2001 Sep;49(9):1205-11. doi: 10.1046/j.1532-5415.2001.49238.x. PMID 11559380
- [Background] Schwartz AR, Bennett ML, Smith PL, De Backer W, Hedner J, Boudewyns A, Van de Heyning P, Ejnell H, Hochban W, Knaack L, Podszus T, Penzel T, Peter JH, Goding GS, Erickson DJ, Testerman R, Ottenhoff F, Eisele DW. Therapeutic electrical stimulation of the hypoglossal nerve in obstructive sleep apnea. Arch Otolaryngol Head Neck Surg. 2001 Oct;127(10):1216-23. doi: 10.1001/archotol.127.10.1216. PMID 11587602
- [Background] Puhan MA, Suarez A, Lo Cascio C, Zahn A, Heitz M, Braendli O. Didgeridoo playing as alternative treatment for obstructive sleep apnoea syndrome: randomised controlled trial. BMJ. 2006 Feb 4;332(7536):266-70. doi: 10.1136/bmj.38705.470590.55. Epub 2005 Dec 23. PMID 16377643
- [Background] Guimaraes KC, Drager LF, Genta PR, Marcondes BF, Lorenzi-Filho G. Effects of oropharyngeal exercises on patients with moderate obstructive sleep apnea syndrome. Am J Respir Crit Care Med. 2009 May 15;179(10):962-6. doi: 10.1164/rccm.200806-981OC. Epub 2009 Feb 20. PMID 19234106